CLINICAL TRIAL: NCT02976818
Title: Relationships Between Lipoprotein(a) Levels and Aortic Valve Calcification in Patients With Heterozygous Familial Hypercholesterolemia
Brief Title: Lp(a) and Aortic Valve Calcification
Acronym: FHLPA
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Patrick Couture, Principal Investigator, Laval University
Other Study IDs: ISS 20167474
Record Dates: First submitted 2016-11-25; First posted 2016-11-29 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Heterozygous Familial Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Aortic valve stenosis (AVS), the most common form of valve disease in the western world, afflicts more than 1 million individuals in North America [1] and the burden of AVS is high and is expected to double within the next 50 years [2]. Medical therapy to prevent development or reduce progression of AVS is currently not available and the only effective treatment for AVS is aortic valve replacement, for which costs have been estimated up to 120,000$ [3,4]. Recently, we and others have identified rs10455872 at the LPA locus as a susceptibility single nucleotide polymorphism (SNP) for aortic valve calcification (AVC) and AVS [5,6] and rs10455872 is associated with elevated plasma lipoprotein (Lp)(a) levels [7]. Lp(a) is a LDL-like particle consisting of hepatically synthesized apolipoprotein B-100 that is noncovalently bound to the plasminogen-like glycoprotein apolipoprotein(a) [8]. Lp(a) promotes atherosclerotic stenosis, and possibly thrombosis, and has been hypothesized to contribute to wound healing, each of which could explain an association with AVS [9,10]. Lp(a) is relatively refractory to both lifestyle and drug intervention, with only nicotinic acid and monoclonal antibody inhibition of the proprotein convertase subtilisin/kexin type 9 that have showed reductions in Lp(a) levels [11,12]. However, the evidence that patients with AVS could be characterized by high Lp(a) levels is scarce. Glader et al. [13] showed that plasma levels of Lp(a) were almost 1.5-fold higher in 101 patients with AVS compared to matched controls, although this relationship did not reach statistical significance. Subsequent studies have also reported an association between elevated plasma Lp(a) levels and higher prevalence of AVS. More specifically, Kamstrup and colleagues [14] reported that elevated Lp(a) levels and corresponding genotypes were associated with increased risk of AVS in the general population with levels >90 mg/dL predicting a threefold increased risk. We have measured Lp(a) and oxidized phospholipids plasma levels in 220 patients with mild-to-moderate calcific AVS enrolled in the Aortic Stenosis Progression Observation: Measuring Effects of Rosuvastatin (ASTRONOMER) trial [15]. Results of this study suggest that high Lp(a) and oxidized phospholipids both predict calcific AVS progression, especially in younger patients with calcific AVS. We also found that statin therapy considerably increased both Lp(a) and oxidized phospholipids levels. Whether the fact that statins increase these risk factors for calcific AVS might explain at least to a certain extent why statins failed to promote calcific AVS regression or stabilization in at least four trials, including ASTRONOMER.

Familial hypercholesterolemia (FH) is an autosomal codominant single-gene disorder caused by mutations in the LDL receptor gene that disrupt normal clearance of LDL. Phenotypic features characteristic of the disease's heterozygous form are 2- to 3-fold raise in plasma LDL-cholesterol concentrations, tendinous xanthomatosis and premature atherosclerotic coronary artery disease. High Lp(a) levels have been shown to explain residual cardiovascular disease risk in FH [16,17]. Recent studies have demonstrated that FH heterozygotes have elevated AVC compared with non-FH subjects [18] and that Lp(a) levels were positively correlated with AVC in asymptomatic FH heterozygotes [19]. Vongpromek et al. [19] demonstrated that plasma Lp(a) concentration is a independent risk factor for AVC in a cohort of 129 asymptomatic heterozygous FH patients aged between 40 and 69 years. In this study, AVC was significantly associated with plasma Lp(a) level, age, body mass index, blood pressure, duration of statin use, cholesterol-year score and coronary artery calcification (CAC) score.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with heterozygous FH aged between 18 and 80 years
* FH patient carrying a documented mutation in the LDL receptor gene
* Subjects must be willing to give written informed consent and able to adhere to visit schedule

Exclusion Criteria:

* Men or women < 18 or > 80 years
* Non-FH subjects
* History of alcohol or drug abuse within the past 2 years
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Association between Lp(a) concentrations and aortic valve calcification | Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, FRCP, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iung B, Vahanian A. Degenerative calcific aortic stenosis: a natural history. Heart. 2012 Nov;98 Suppl 4:iv7-13. doi: 10.1136/heartjnl-2012-302395. PMID 23143128
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jun 10;63(22):2438-88. doi: 10.1016/j.jacc.2014.02.537. Epub 2014 Mar 3. No abstract available. PMID 24603192
- [Background] Utermann G. The mysteries of lipoprotein(a). Science. 1989 Nov 17;246(4932):904-10. doi: 10.1126/science.2530631.
- [Result] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Result] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Result] Thanassoulis G, Campbell CY, Owens DS, Smith JG, Smith AV, Peloso GM, Kerr KF, Pechlivanis S, Budoff MJ, Harris TB, Malhotra R, O'Brien KD, Kamstrup PR, Nordestgaard BG, Tybjaerg-Hansen A, Allison MA, Aspelund T, Criqui MH, Heckbert SR, Hwang SJ, Liu Y, Sjogren M, van der Pals J, Kalsch H, Muhleisen TW, Nothen MM, Cupples LA, Caslake M, Di Angelantonio E, Danesh J, Rotter JI, Sigurdsson S, Wong Q, Erbel R, Kathiresan S, Melander O, Gudnason V, O'Donnell CJ, Post WS; CHARGE Extracoronary Calcium Working Group. Genetic associations with valvular calcification and aortic stenosis. N Engl J Med. 2013 Feb 7;368(6):503-12. doi: 10.1056/NEJMoa1109034. PMID 23388002
- [Result] Arsenault BJ, Boekholdt SM, Dube MP, Rheaume E, Wareham NJ, Khaw KT, Sandhu MS, Tardif JC. Lipoprotein(a) levels, genotype, and incident aortic valve stenosis: a prospective Mendelian randomization study and replication in a case-control cohort. Circ Cardiovasc Genet. 2014 Jun;7(3):304-10. doi: 10.1161/CIRCGENETICS.113.000400. Epub 2014 Apr 5. PMID 24704946
- [Result] Clarke R, Peden JF, Hopewell JC, Kyriakou T, Goel A, Heath SC, Parish S, Barlera S, Franzosi MG, Rust S, Bennett D, Silveira A, Malarstig A, Green FR, Lathrop M, Gigante B, Leander K, de Faire U, Seedorf U, Hamsten A, Collins R, Watkins H, Farrall M; PROCARDIS Consortium. Genetic variants associated with Lp(a) lipoprotein level and coronary disease. N Engl J Med. 2009 Dec 24;361(26):2518-28. doi: 10.1056/NEJMoa0902604. PMID 20032323
- [Result] Helgadottir A, Gretarsdottir S, Thorleifsson G, Holm H, Patel RS, Gudnason T, Jones GT, van Rij AM, Eapen DJ, Baas AF, Tregouet DA, Morange PE, Emmerich J, Lindblad B, Gottsater A, Kiemeny LA, Lindholt JS, Sakalihasan N, Ferrell RE, Carey DJ, Elmore JR, Tsao PS, Grarup N, Jorgensen T, Witte DR, Hansen T, Pedersen O, Pola R, Gaetani E, Magnadottir HB, Wijmenga C, Tromp G, Ronkainen A, Ruigrok YM, Blankensteijn JD, Mueller T, Wells PS, Corral J, Soria JM, Souto JC, Peden JF, Jalilzadeh S, Mayosi BM, Keavney B, Strawbridge RJ, Sabater-Lleal M, Gertow K, Baldassarre D, Nyyssonen K, Rauramaa R, Smit AJ, Mannarino E, Giral P, Tremoli E, de Faire U, Humphries SE, Hamsten A, Haraldsdottir V, Olafsson I, Magnusson MK, Samani NJ, Levey AI, Markus HS, Kostulas K, Dichgans M, Berger K, Kuhlenbaumer G, Ringelstein EB, Stoll M, Seedorf U, Rothwell PM, Powell JT, Kuivaniemi H, Onundarson PT, Valdimarsson E, Matthiasson SE, Gudbjartsson DF, Thorgeirsson G, Quyyumi AA, Watkins H, Farrall M, Thorsteinsdottir U, Stefansson K. Apolipoprotein(a) genetic sequence variants associated with systemic atherosclerosis and coronary atherosclerotic burden but not with venous thromboembolism. J Am Coll Cardiol. 2012 Aug 21;60(8):722-9. doi: 10.1016/j.jacc.2012.01.078. PMID 22898070
- [Result] Yano Y, Shimokawa K, Okada Y, Noma A. Immunolocalization of lipoprotein(a) in wounded tissues. J Histochem Cytochem. 1997 Apr;45(4):559-68. doi: 10.1177/002215549704500408. PMID 9111234
- [Result] AIM-HIGH Investigators; Boden WE, Probstfield JL, Anderson T, Chaitman BR, Desvignes-Nickens P, Koprowicz K, McBride R, Teo K, Weintraub W. Niacin in patients with low HDL cholesterol levels receiving intensive statin therapy. N Engl J Med. 2011 Dec 15;365(24):2255-67. doi: 10.1056/NEJMoa1107579. Epub 2011 Nov 15. PMID 22085343
- [Result] Raal F, Scott R, Somaratne R, Bridges I, Li G, Wasserman SM, Stein EA. Low-density lipoprotein cholesterol-lowering effects of AMG 145, a monoclonal antibody to proprotein convertase subtilisin/kexin type 9 serine protease in patients with heterozygous familial hypercholesterolemia: the Reduction of LDL-C with PCSK9 Inhibition in Heterozygous Familial Hypercholesterolemia Disorder (RUTHERFORD) randomized trial. Circulation. 2012 Nov 13;126(20):2408-17. doi: 10.1161/CIRCULATIONAHA.112.144055. Epub 2012 Nov 5. PMID 23129602
- [Result] Glader CA, Birgander LS, Soderberg S, Ildgruben HP, Saikku P, Waldenstrom A, Dahlen GH. Lipoprotein(a), Chlamydia pneumoniae, leptin and tissue plasminogen activator as risk markers for valvular aortic stenosis. Eur Heart J. 2003 Jan;24(2):198-208. doi: 10.1016/s0195-668x(02)00385-8. PMID 12573277
- [Result] Kamstrup PR, Tybjaerg-Hansen A, Nordestgaard BG. Elevated lipoprotein(a) and risk of aortic valve stenosis in the general population. J Am Coll Cardiol. 2014 Feb 11;63(5):470-7. doi: 10.1016/j.jacc.2013.09.038. Epub 2013 Oct 23. PMID 24161338
- [Result] Capoulade R, Chan KL, Yeang C, Mathieu P, Bosse Y, Dumesnil JG, Tam JW, Teo KK, Mahmut A, Yang X, Witztum JL, Arsenault BJ, Despres JP, Pibarot P, Tsimikas S. Oxidized Phospholipids, Lipoprotein(a), and Progression of Calcific Aortic Valve Stenosis. J Am Coll Cardiol. 2015 Sep 15;66(11):1236-1246. doi: 10.1016/j.jacc.2015.07.020. PMID 26361154
- [Result] Jansen AC, van Aalst-Cohen ES, Tanck MW, Trip MD, Lansberg PJ, Liem AH, van Lennep HW, Sijbrands EJ, Kastelein JJ. The contribution of classical risk factors to cardiovascular disease in familial hypercholesterolaemia: data in 2400 patients. J Intern Med. 2004 Dec;256(6):482-90. doi: 10.1111/j.1365-2796.2004.01405.x. PMID 15554949
- [Result] Seed M, Hoppichler F, Reaveley D, McCarthy S, Thompson GR, Boerwinkle E, Utermann G. Relation of serum lipoprotein(a) concentration and apolipoprotein(a) phenotype to coronary heart disease in patients with familial hypercholesterolemia. N Engl J Med. 1990 May 24;322(21):1494-9. doi: 10.1056/NEJM199005243222104. PMID 2139920
- [Result] Ten Kate GR, Bos S, Dedic A, Neefjes LA, Kurata A, Langendonk JG, Liem A, Moelker A, Krestin GP, de Feyter PJ, Roeters van Lennep JE, Nieman K, Sijbrands EJ. Increased Aortic Valve Calcification in Familial Hypercholesterolemia: Prevalence, Extent, and Associated Risk Factors. J Am Coll Cardiol. 2015 Dec 22;66(24):2687-2695. doi: 10.1016/j.jacc.2015.09.087. PMID 26700830
- [Result] Vongpromek R, Bos S, Ten Kate GJ, Yahya R, Verhoeven AJ, de Feyter PJ, Kronenberg F, Roeters van Lennep JE, Sijbrands EJ, Mulder MT. Lipoprotein(a) levels are associated with aortic valve calcification in asymptomatic patients with familial hypercholesterolaemia. J Intern Med. 2015 Aug;278(2):166-73. doi: 10.1111/joim.12335. Epub 2015 Jan 5. PMID 25487646